CLINICAL TRIAL: NCT04265937
Title: Screening of Genetic Susceptibility Genes for Breast Cancer Patients and Establishment of High-risk Populations in Chinese Communities
Brief Title: ScreenIng of Genetic Susceptibility Genes for Breast Cancer Patients in CHinese communiTies
Acronym: SIGHT
Status: Recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhen Hu, Professor, Fudan University
Other Study IDs: 1905202-3
Record Dates: First submitted 2020-02-08; First posted 2020-02-12 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Breast Cancer; Genetic Susceptibility
MeSH Terms: conditions — Breast Neoplasms; Genetic Predisposition to Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood or oral mucosa samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a community-based prospective study and the research object is breast cancer patients. It is planned to take the community as the unit to inform and collect the breast cancer patients who voluntarily participate to carry out the detection of BRCA1, BRCA2, PTEN, CHEK2 and PALB2 genes through the community health service center.

DETAILED DESCRIPTION:
This is a population-based, prospective, cohort study which has been ongoing in 3 provinces of eastern China since 2019. Up to 5000 breast cancer survivors will conduct BRCA1, BRCA2, PTEN, CHEK2, and PALB2 genetic susceptibility genes testing, fill in clinical and genetic information forms, and collect family history. Mutation rate of BRCA1/2 and other genetic susceptibility genes in Chinese community breast cancer population will be measured. Logistic regression will be performed to establish a prediction model for the probability of BRCA1/2 and other gene mutations. Kin-Cohort method will be used to calculate the penetrance of breast cancer and other common malignancies in BRCA1/2 and other genetic mutation carriers.

ELIGIBILITY:
Inclusion Criteria:

* breast cancer patients of any age;
* both male and female;
* the subjects signed the informed consent to participate in the study and abide by the study procedure before being selected.

Exclusion Criteria:

* healthy people or other malignant tumor patients without breast cancer;
* unable to interview the investigator and sign the informed consent due to any reason;
* it is impossible to collect peripheral blood or oral mucosa samples for any reason.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Breast cancer patients from community.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
The frequency of pathogenic or likely pathogenic variants of BRCA1/2 and other genetic susceptibility genes in Chinese community breast cancer population | 1 year
  The frequency of pathogenic or likely pathogenic variants and 95% confidence intervals of BRCA1/2 and other genetic susceptibility genes in Chinese community breast cancer population will be measured. After stratifying according to the different clinical characteristics of the patients, chi-square tests will be use to compare the mutation rates of BRCA1/2 gene in different subgroups.

SECONDARY OUTCOMES:
Prediction model of Genetic Susceptibility Gene (BRCA1/2 etc) mutation probability | 1 year
  Logistic regression will be performed to establish a prediction model for the probability of pathogenic or likely pathogenic variants of BRCA1/2 and other genes. Candidate predictors included age, race or ethnic group, the mean number of tumor in a family etc. Missing data were imputed using multiple imputation by chained equations if needed. Model validation is based on k-fold cross validation approach. Model calibration and discrimination were evaluated using HL test and AUC, respectively. ORs and corresponding 95% CI will report.
Breast cancer penetrance of Genetic Susceptibility Gene (BRCA1/2 etc) carriers | 1 year
  Kin-Cohort method will be used to calculate the penetrance of breast cancer and other common malignancies in BRCA1/2 and other genetic mutation carriers.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhen Hu, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Yu S, Qiu X, Wang Z, Xiao J, Ji H, Shan H, Shao Q, Xia H, Cao F, Li J, Fu C, Chen L, Lu X, Su T, Yu Q, Hou S, Wang H, Zheng Y, Shao Z, Liu Y, Hu Z. Breast cancer risk associated with BRCA1 and BRCA2 pathogenic variants in the Eastern Chinese population. Cancer Pathog Ther. 2024 Apr 17;3(2):147-153. doi: 10.1016/j.cpt.2024.04.002. eCollection 2025 Mar. PMID 40182128